CLINICAL TRIAL: NCT06983899
Title: Boosting the Effects of Immunotherapy Through Exercise Training in Patients With Lung Cancer: The BOOST Trial
Brief Title: Exercise Training for the Improvement of Immune Activity and Treatment Outcomes During Immunotherapy for Non-small Cell Lung Cancer, BOOST Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1125289; NCI-2025-02781 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20819 (Other: Fred Hutch/University of Washington Cancer Consortium); R00CA287050 (NIH)
Record Dates: First submitted 2025-04-30; First posted 2025-05-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Exercise; Early Intervention, Educational; Educational Status; Methods; Absorptiometry, Photon; Bone Density; Exercise Test; Clostridium perfringens epsilon-toxin; Respiratory Physiological Phenomena

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (aerobic training sessions, equipment, guidebook) (Experimental): Patients complete virtual home-based aerobic interval training sessions with a trained exercise specialist via stationary bike over approximately 60 minutes QW during weeks 1-4, BIW during weeks 5-8, and TIW during weeks 9-24 in the absence of unacceptable toxicity. Patients also receive a stationary bike, HR monitor, BP monitor, SPO2 monitor, and a general healthy lifestyle guidebook for cancer patients and survivors on study. Patients also undergo blood sample collection, dual-energy x-ray absorptiometry (DEXA), pulmonary function test (PFT), physical fitness and function tests, and questionnaires throughout the study.
  Interventions: Other: Aerobic Exercise; Other: Exercise Intervention; Other: Educational Intervention; Procedure: Dual X-ray Absorptiometry; Other: Electronic Health Record Review; Other: Cardiopulmonary Exercise Testing; Other: Physical Performance Testing; Other: Questionnaire Administration; Procedure: Biospecimen Collection; Procedure: Pulmonary Function Test
- Arm II (guidebook) (Active Comparator): Patients receive a general healthy lifestyle guidebook for cancer patients and survivors on study. Patients also undergo blood sample collection, dual-energy x-ray absorptiometry (DEXA), pulmonary function test (PFT), physical fitness and function tests, and questionnaires throughout the study.
  Interventions: Other: Educational Intervention; Procedure: Dual X-ray Absorptiometry; Other: Electronic Health Record Review; Other: Cardiopulmonary Exercise Testing; Other: Physical Performance Testing; Other: Questionnaire Administration; Procedure: Biospecimen Collection; Procedure: Pulmonary Function Test

INTERVENTIONS:
Other: Aerobic Exercise — Complete virtual home-based aerobic interval training sessions
  Other Names: Aerobic Activity
  Arms: Arm I (aerobic training sessions, equipment, guidebook)
Other: Exercise Intervention — Receive stationary bike, HR monitor, BP monitor, SPO2 monitor
  Arms: Arm I (aerobic training sessions, equipment, guidebook)
Other: Educational Intervention — Receive general healthy lifestyle guidebook
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Procedure: Dual X-ray Absorptiometry — Undergo DEXA
  Other Names: BMD scan; bone mineral density scan; DEXA; DEXA (Bone Density); DEXA Scan; dual energy x-ray absorptiometric scan; Dual Energy X-ray Absorptiometry; Dual X-Ray Absorptometry; DXA; DXA SCAN
Other: Electronic Health Record Review — Ancillary studies
Other: Cardiopulmonary Exercise Testing — Ancillary studies
  Other Names: CPET; CPX
Other: Physical Performance Testing — Ancillary studies
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Questionnaire Administration — Ancillary studies
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection
Procedure: Pulmonary Function Test — Undergo PFT
  Other Names: PFT

SUMMARY:
This clinical trial studies how well exercise training works in improving immune activity and treatment tolerance and response in patients with non-small cell lung cancer (NSCLC) who are receiving immunotherapy. Immunotherapy may induce changes in the body's immune system and may interfere with the ability of tumor cells to grow and spread. The use of immunotherapy for the treatment of NSCLC has been rapidly increasing. Although immunotherapy have shown great potential in cancer therapy, not all patients benefit from this therapy and resistance to it can occur. This could be due to poor immune activity. It has been shown that exercise can enhance systemic immune activity in various ways. The exercise training used in this study is aerobic interval training. Aerobic interval training increases the heart rate and the body's use of oxygen and alternates short periods of intense aerobic exercise with less intense recovery periods. This may cause biological changes which may improve immune activity and treatment response in patients with NSCLC who are receiving immunotherapy.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients complete virtual home-based aerobic interval training sessions with a trained exercise specialist via stationary bike over approximately 60 minutes once a week (QW) during weeks 1-4, twice a week (BIW) during weeks 5-8, and three times a week (TIW) during weeks 9-24 in the absence of unacceptable toxicity. Patients also receive a stationary bike, heart rate (HR) monitor, blood pressure (BP) monitor, oxygen saturation (SPO2) monitor, and a general healthy lifestyle guidebook for cancer patients and survivors on study. Patients also undergo blood sample collection, dual-energy x-ray absorptiometry (DEXA), pulmonary function test (PFT), physical fitness and function tests, and questionnaires throughout the study.

ARM II: Patients receive a general healthy lifestyle guidebook for cancer patients and survivors on study. Patients also undergo blood sample collection, DEXA, PFT, physical fitness and function tests, and questionnaires throughout the study.

After completion of study intervention, patients are followed up at week 26 and then every 3 months up to the completion of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically diagnosed with NSCLC.
* Currently receiving immunotherapy with a minimum of one month of treatment completed.
* Having a plan to continue immunotherapy for at least 24 weeks (i.e., study intervention period) at the time of recruitment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2, indicating the ability to fulfill physical fitness and function assessments.
* Able to understand and willingness to provide study consent.

Exclusion Criteria:

* Participating in ≥ 150 minutes of moderate-to-vigorous aerobic exercise per week over the past month. This study targets insufficiently active persons to assess the effect of the described exercise intervention, where additional exercise done regularly will contaminate the intervention outcomes.
* Having medical conditions clinically unstable or uncontrollable, with medications that are deemed high-risk for exercise participation by the study team in consultation with the treating oncologist, using the electric medical record (EMR) and Physical Activity Readiness Questionnaire (PAR-Q). This includes but is not limited to: recent (< 6 months) myocardial infarction, uncontrolled arrhythmias, decompensated heart failure, unstable angina, symptomatic severe aortic stenosis, uncontrolled hypertension (≥ 180/110 mmHg), uncontrolled diabetes (hemoglobin A1c [HbA1c] > 10% with symptoms), severe chronic obstructive pulmonary disease requiring hospitalization in past 3 months, and bone metastases with imminent fracture risk. These exclusions are based on the American College of Sports Medicine (ACSM)'s Guidelines for Exercise Testing and Prescription and the American Association of Cardiovascular and Pulmonary Rehabilitation (AACPR)'s Guidelines for Cardiac Rehabilitation Programs for safe exercise in clinical populations.
* Having a high risk for noncompliance with study procedures, including but not limited to: informed consent, participation in outcome assessments, completion of fasting blood draws, attendance at scheduled sessions, adherence to supervised virtual exercise sessions, and appropriate use of provided monitoring equipment (e.g., heart rate monitor, blood pressure monitor, SpO2 monitor). This determination will be based on a composite assessment of the following factors: history of missed oncology appointments (i.e., three or more uninformed no-shows in the prior six months) and poor responsiveness to study communications (i.e., three or more repeated unreturned calls or emails during the recruitment stage). We will also consider any demonstrated difficulty following instructions during initial scheduling or onboarding, or clinical concern raised by the referring provider. Participants meeting one or more of these criteria likely to impair participation will be considered ineligible.
* Patients who are non-English speaking that would prevent their participation in the participant survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Mean difference in neutrophil-to-lymphocyte ratio (NLR) | Baseline (Week 1) and post-intervention (Week 26)
  The primary analysis will follow an intention-to-treat approach, using a two-sample t-test to compare changes in NLR from baseline between the groups.

SECONDARY OUTCOMES:
Mean difference in immune parameters | Baseline (Week 1) and post-intervention (Week 26)
  To analyze changes in immune parameters (e.g., T-cells, natural killer cells, B-cells) a two-sample t-test will compare changes between the groups.
Mean difference in inflammatory cytokines | Baseline (Week 1) and post-intervention (Week 26)
  To analyze changes in inflammatory cytokines (e.g., IL-6, IL-15) a two-sample t-test will compare changes between the groups.
Mean change in fasting glucose (mg/dL) | Baseline (Week 1) and post-intervention (Week 26)
Mean change in insulin (µIU/mL) | Baseline (Week 1) and post-intervention (Week 26)
Mean change in lipid profile | Baseline (Week 1) and post-intervention (Week 26)
Mean difference in circulating tumor markers | Baseline (Week 1) and post-intervention (Week 26)
  To analyze changes in tumor markers [e.g., circulating tumor deoxyribonucleic acid (DNA)] a two-sample t-test will compare changes between the groups.
Mean change in body weight (kg), assessed via weight scale | Baseline (Week 1) and post-intervention (Week 26)
Mean change in body mass index (BMI) (kg/m²), calculated from height and weight | Baseline (Week 1) and post-intervention (Week 26)
Mean change in lean mass (kg), assessed via DEXA | Baseline (Week 1) and post-intervention (Week 26)
Mean change in body fat percentage (%), assessed via DEXA | Baseline (Week 1) and post-intervention (Week 26)
Mean change in body fat mass (kg), assessed via DEXA | Baseline (Week 1) and post-intervention (Week 26)
Mean change in FEV (L), assessed via spirometry | Baseline (Week 1) and post-intervention (Week 26)
Mean change in FEV1 (L), derived from FEV1 | Baseline (Week 1) and post-intervention (Week 26)
Mean change in FEV1/FEV, derived from FEV and FEV1A | Baseline (Week 1) and post-intervention (Week 26)
Mean difference in cardiopulmonary fitness | Baseline (Week 1) and post-intervention (Week 26)
  Will be assessed as peak oxygen consumption (VO2peak) by a graded maximal or submaximal cycle exercise stress test. VO2peak is defined as the highest values of oxygen uptake averaged over set intervals (i.e., 30-second) during the test. VO2peak will be reported in both relative and absolute terms.
Mean difference in timed balance | Baseline (Week 1) and post-intervention (Week 26)
  Balance will be assessed under 3 conditions: a) side-by-side stand with both feet plated on the ground for 10 seconds or when the subject steps out of position; b) semi-tandem stand with the side of the heel of one foot touching the big toe of the other foot for 10 seconds or when the subject steps out of position; c) tandem stand with the heel of one foot touching the big toe of the other foot for 10 seconds or when the subject steps out of position.
Mean difference in gait speed | Baseline (Week 1) and post-intervention (Week 26)
  Gait speed will be assessed over a 4-meter flat surface distance. The participant will be asked to complete 2 attempts of this test. Time will be recorded using an electronic timing system.
Mean difference in chair stand | Baseline (Week 1) and post-intervention (Week 26)
  Chair stand will be assessed that subjects will perform a single chair stand and if successful, they will be asked to perform 5 repeated chair stands as quickly as possible; time to completion will be recorded.
Mean difference in health-related quality of life | Baseline (Week 1) and post-intervention (Week 26)
  Health-related quality of life will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30. The scale ranges from 0 to 100, with higher scores on the global health status and functioning scales indicating better quality of life, and higher scores on symptom scales indicating worse symptoms.
Mean difference in lung cancer-related quality of life | Baseline (Week 1) and post-intervention (Week 26)
  Lung cancer-related quality of life will be assessed at baseline and post-intervention using the EORTC QLQ-Lung Cancer 29 (QLQ-LC29). The scale ranges from 0 to 100, with higher functioning scores indicating better quality of life and higher symptom scores indicating worse symptoms.
Mean difference in immunotherapy-related symptoms | Baseline (Week 1), mid-point (Week 13), post-intervention (Week 26), and every three months post-intervention up to the completion of immunotherapy.
  Immunotherapy-related symptoms will be assessed at baseline, mid-point, post-intervention, and during follow-up using the MD Anderson Symptom Inventory (MDASI) Immunotherapy Early Phase Trials module (EPT). Each symptom is rated from 0 ("not present") to 10 ("as bad as you can imagine"), with higher scores indicating worse symptom severity.
Mean difference in symptomatic treatment toxicity | Baseline (Week 1), mid-point (Week 13), post-intervention (Week 26), and every three months post-intervention up to the completion of immunotherapy.
  Symptomatic treatment toxicity will be assessed at baseline, mid-point, post-intervention, and during follow-up using the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). Each item is rated from 0 to 4, with higher scores indicating greater severity, frequency, or interference of adverse events.
Mean difference in anxiety and depression | Baseline (Week 1) and post-intervention (Week 26)
  Will be assessed using the Hospital Anxiety and Depression Scale. Each subscale (anxiety and depression) ranges from 0 to 21, with higher scores indicating greater levels of anxiety or depression.
Mean difference in sleep quality | Baseline (Week 1) and post-intervention (Week 26)
  Will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The global PSQI score ranges from 0 to 21, with higher scores indicating poorer sleep quality.
Mean difference in exercise behavior | Baseline (Week 1), mid-point (Week 13), post-intervention (Week 26), and every three months post-intervention up to the completion of immunotherapy.
  Exercise behavior will be assessed at baseline, mid-point, post-intervention, and during follow-up using the Godin Leisure-Time Exercise Questionnaire (GLTEQ). Weekly exercise scores are calculated, with higher scores indicating greater amounts of physical activity. A minimum value is 0 and maximum value is 10080 minutes per week.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Woo Kang, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No